CLINICAL TRIAL: NCT00944190
Title: Telephone Delivered Self-management Intervention for People With Multiple Sclerosis Addressing Pain, Fatigue, Depression, and Cognitive Difficulties
Brief Title: TakeCharge: Telephone Delivered Self-management Intervention for People With Multiple Sclerosis (MS)
Acronym: TakeCharge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Dawn Ehde, Professor, Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36021-C; H133B080025 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis
Keywords: pain; fatigue; depression; cognitive difficulties; self-management
MeSH Terms: conditions — Multiple Sclerosis; Pain; Fatigue; Depression | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-management Intervention (Experimental): Telephone based self management intervention targeted at pain, fatigue, depression, and cognitive difficulties.
  Interventions: Behavioral: Self-management intervention
- Education (Active Comparator): Education about pain, fatigue, depression, and cognitive difficulties in multiple sclerosis.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Self-management intervention — Brief counseling technique, self-management,
  Arms: Self-management Intervention
Behavioral: Education — Educational information about pain, fatigue, depression, and cognitive difficulties in multiple sclerosis.
  Arms: Education

SUMMARY:
The proposed project will evaluate the efficacy of a telephone-delivered self-management (T-SM) intervention for reducing the impact of secondary conditions in persons with multiple sclerosis (MS), including chronic pain, fatigue, depression, and cognitive impairment. It is hypothesized that if the effects of these conditions are reduced, study participants will demonstrate improved participation in the community and improved employment outcomes. This project is important because the majority of persons with MS experience one or more of the following secondary conditions: fatigue, pain, depression, and cognitive impairment. These secondary conditions are not always readily apparent and constitute what has been described by our Rehabilitation Research and Training Center as "hidden disabilities." Secondary conditions such as pain, depression, fatigue, and cognitive impairment frequently not only cause distress in their own right but also affect employment, participation, and quality of life. Having more than one often compounds the effect; the effect of all may be greater than the sum of each individually (e.g. depression can worsen fatigue, and cognitive impairment can worsen depression).

It is critical that this constellation of secondary symptoms be addressed using state of the art techniques based on self-management training and that intervention effects be documented with carefully controlled treatment efficacy studies.

ELIGIBILITY:
Inclusion Criteria:

* Must be diagnosed with MS by a physician.
* Must be at least 18 years of age.
* Must be able to understand, speak, and read English.
* Must have the presence of at least one of four common secondary conditions (fatigue, pain, depression, cognitive difficulties) that interferes with employment, participation, and functioning.

Exclusion Criteria:

* Unable to understand or read English.
* Severe cognitive impairment, defined as one or more errors on the 6-item screener, that would prevent informed consent and inability to carry on a phone conversation.
* Currently participating in regularly scheduled psychotherapy.
* Psychiatric contraindications such as current psychosis, active suicidal ideation, or current alcohol or drug use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
PHQ 9 | Baseline, 5 weeks, 10 weeks, 6 months, and 12 months
Brief Pain Inventory | Baseline, 5 weeks, 10 weeks, 6 months, and 12 months
Modified Fatigue Impact Scale | Baseline, 5 weeks, 10 weeks, 6 months, 12 months

SECONDARY OUTCOMES:
PROMIS Depression Short Form | Baseline, 5 weeks, 10 weeks, 6 months, 12 months
PROMIS Pain Impact Short Form | Baseline, 5 weeks, 10 weeks, 6 months, 12 months
PROMIS Fatigue Short Form | Baseline, 5 weeks, 10 weeks, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Ehde, PhD, Principal Investigator — University of Washington; George Kraft, MD, Study Director — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Knowles LM, Arewasikporn A, Kratz AL, Turner AP, Alschuler KN, Ehde DM. Early Treatment Improvements in Depression Are Associated With Overall Improvements in Fatigue Impact and Pain Interference in Adults With Multiple Sclerosis. Ann Behav Med. 2021 Aug 23;55(9):833-843. doi: 10.1093/abm/kaaa102. PMID 33196779
- [Derived] Ehde DM, Arewasikporn A, Alschuler KN, Hughes AJ, Turner AP. Moderators of Treatment Outcomes After Telehealth Self-Management and Education in Adults With Multiple Sclerosis: A Secondary Analysis of a Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Jul;99(7):1265-1272. doi: 10.1016/j.apmr.2017.12.012. Epub 2018 Jan 11. PMID 29337024
- [Derived] Ehde DM, Elzea JL, Verrall AM, Gibbons LE, Smith AE, Amtmann D. Efficacy of a Telephone-Delivered Self-Management Intervention for Persons With Multiple Sclerosis: A Randomized Controlled Trial With a One-Year Follow-Up. Arch Phys Med Rehabil. 2015 Nov;96(11):1945-58.e2. doi: 10.1016/j.apmr.2015.07.015. Epub 2015 Aug 6. PMID 26254948
- See also: Webpage for MS Rehabilitation Research and Training Center — http://msrrtc.washington.edu